CLINICAL TRIAL: NCT04915040
Title: Management of Depression and Social Isolation in Older Adults With Dementia With Home-based Telehealth Delivered Behavioral Activation + Caregiver Facilitation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Michael Bradley Cannell, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SPH-21-0272
Record Dates: First submitted 2021-05-31; First posted 2021-06-07 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Depression
Keywords: social support; dementia; caregivers
MeSH Terms: conditions — Depression; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Activation for Depression (Experimental)
  Interventions: Behavioral: Behavioral Activation for Depression

INTERVENTIONS:
Behavioral: Behavioral Activation for Depression — Behavioral Activation (BA) is an effective treatment for depression, and its components may increase social connection. Generally, caregivers are with the older adult care recipient on a regular basis and may be able, with the correct training, to help enhance certain features of the Behavioral Activation treatment, even under pandemic restrictions on social contact. Therefore, we propose to (a) integrate & (b) gather feasibility data for home-based Behavioral Activation + Caregiver

SUMMARY:
The purpose of this study is to evaluate the feasibility of using behavioral activation therapy with caregiver support delivered via telemedicine to older adults with depression and probable mild dementia.

ELIGIBILITY:
Inclusion Criteria:

Participant Eligibility Criteria:

* able to speak and understand English;
* a diagnosis of mild dementia, as determined by a Clinical Dementia Rating interview Sum of Boxes (CDR-SB) score in the mild range as defined by a score of 4.5 - 9.0;
* and able to provide informed consent.

Caregiver Eligibility Criteria.

* Beck Depression Inventory (BDI) score below clinical cutoff for depression and able to provide informed consent.

Exclusion Criteria:

Participant exclusion criteria:

* presence of suicidal ideation with clear intent,
* concurrent enrollment in another clinical trial for depression,
* substance use disorder.

Caregiver exclusion criteria:

* Active psychosis or significant dementia at screening;
* presence of suicidal ideation with clear intent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment as assessed by number of participants enrolled in the study | Week 0
Feasibility of retention as assessed by number of participants who complete at least 6 sessions | Week 8
Feasibility of data collection as assessed by percent of missing data | Week 8
Change in Depression as measured by the Geriatric Depression Scale | Week 0, Week 4, Week 8
  15-item self-report for each construct (yes/no) . Score goes from 1 to 15, a higher number indicates presence of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No